CLINICAL TRIAL: NCT03206580
Title: Functional Mobility in the Elderly: Influence of Morphological, Neuromuscular and Training
Brief Title: Functional Mobility in the Elderly: Influence of Morphological, Neuromuscular and Training Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Marco Aurélio Vaz, PhD, Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UFRGS 2.034.508
Record Dates: First submitted 2017-06-22; First posted 2017-07-02 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Aging
Keywords: aging; strength training; functionality

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concentric training (Experimental): Concentric training
  Interventions: Other: Concentric training
- Concentric-eccentric training (Experimental): Concentric-eccentric training
  Interventions: Other: Concentric-Eccentric training

INTERVENTIONS:
Other: Concentric training — Subjects will be submitted to 8 weeks (16 sessions) of a concentric training for knee flexors and knee extensors. This training will be performed in an isokinetic dynamometer at 70% of the subject's maximal voluntary isometric contraction.
  Arms: Concentric training
Other: Concentric-Eccentric training — Subjects will be submitted to 8 weeks (16 sessions) of a concentric-eccentric training for knee flexors and knee extensors. This training will be performed in an isokinetic dynamometer at 70% of the subject's maximal voluntary isometric contraction.
  Arms: Concentric-eccentric training

SUMMARY:
Life expectancy and elderly population are increasing. Health professionals try to provide longevity with good quality of life for this population, through the functional independence maintenance. In this context, physical exercise has an important role, specially the strength training. The ability to produce muscle strength is positively associated with the functionality and independence of older people. Different types of strength training can lead to different neuromuscular and functional gains. These types of interventions can help health professionals to determine characteristics of training for the elderly, aiming the maintenance of their functional independence. Thus, the purpose of this study is to determine the effects of a concentric strength training versus a concentric-eccentric strength training for knee flexors and extensors on structural, neuromuscular and functional parameters in older people, as well as to investigate the effect of a detraining period. Additionally, the investigators will try to identify which structural and neuromuscular parameters of lower limbs are better related to the functionality.

ELIGIBILITY:
Inclusion Criteria:

* Male;
* 65 years of age or more;
* able to walk independently;
* not engaged in regular physical exercise.

Exclusion Criteria:

* Auditory, vestibular, visual and/or neuromusculoskeletal impairments that could influence the tests and the training;
* severe cognitive impairment;
* lower limb surgery;
* osteoporosis;
* lower limb pain.

Ages: 65 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-10-15 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Pennation angle of rectus femoris, vastus lateralis and biceps femoris, bilaterally. | First evaluation, change from first evaluation to baseline, change from baseline to 8 weeks of training, change from 8 weeks of training to 4 weeks of detraining and change from 4 weeks of detraining to 8 weeks of detraining
  Pennation angle at rest
Thickness of rectus femoris, vastus lateralis and biceps femoris, bilaterally. | First evaluation, change from first evaluation to baseline, change from baseline to 8 weeks of training, change from 8 weeks of training to 4 weeks of detraining and change from 4 weeks of detraining to 8 weeks of detraining
  Muscle thickness at rest
Fascicle length of rectus femoris, vastus lateralis and biceps femoris, bilaterally. | First evaluation, change from first evaluation to baseline, change from baseline to 8 weeks of training, change from 8 weeks of training to 4 weeks of detraining and change from 4 weeks of detraining to 8 weeks of detraining
  Fascicle length at rest
Echo intensity of rectus femoris, vastus lateralis and biceps femoris, bilaterally. | First evaluation, change from first evaluation to baseline, change from baseline to 8 weeks of training, change from 8 weeks of training to 4 weeks of detraining and change from 4 weeks of detraining to 8 weeks of detraining
  Echo intensity determined from a gray scale analysis of the muscles at rest
Countermovement vertical jump | First evaluation, change from first evaluation to baseline, change from baseline to 8 weeks of training, change from 8 weeks of training to 4 weeks of detraining and change from 4 weeks of detraining to 8 weeks of detraining
  Maximal vertical height in the countermovement jump
Timed-up-&-go | First evaluation, change from first evaluation to baseline, change from baseline to 8 weeks of training, change from 8 weeks of training to 4 weeks of detraining and change from 4 weeks of detraining to 8 weeks of detraining
  Time to rise from a chair, walk 3 meters, turn, walk back and sit again
Unipodal static balance | First evaluation, change from first evaluation to baseline, change from baseline to 8 weeks of training, change from 8 weeks of training to 4 weeks of detraining and change from 4 weeks of detraining to 8 weeks of detraining
  Range in anterior-posterior and medio-lateral center of pressure movement during unipodal evaluation during 30 seconds
Gait speed | First evaluation, change from first evaluation to baseline, change from baseline to 8 weeks of training, change from 8 weeks of training to 4 weeks of detraining and change from 4 weeks of detraining to 8 weeks of detraining
  Gait speed for walking 10 meters at self-selected speed
Stair ascent and descent time | First evaluation, change from first evaluation to baseline, change from baseline to 8 weeks of training, change from 8 weeks of training to 4 weeks of detraining and change from 4 weeks of detraining to 8 weeks of detraining
  Time to stair ascent and descent stairs
6-minutes walking test | First evaluation, change from first evaluation to baseline, change from baseline to 8 weeks of training, change from 8 weeks of training to 4 weeks of detraining and change from 4 weeks of detraining to 8 weeks of detraining
  The distance that the subjects can walk during 6 minutes
Sit-to-stand | First evaluation, change from first evaluation to baseline, change from baseline to 8 weeks of training, change from 8 weeks of training to 4 weeks of detraining and change from 4 weeks of detraining to 8 weeks of detraining
  Maximal number of repetitions during 30 seconds
Power of knee extensors and knee flexors | First evaluation, change from first evaluation to baseline, change from baseline to 8 weeks of training, change from 8 weeks of training to 4 weeks of detraining and change from 4 weeks of detraining to 8 weeks of detraining
  Power during maximal concentric and eccentric contractions
Rate of torque production of knee extensors and knee flexors | First evaluation, change from first evaluation to baseline, change from baseline to 8 weeks of training, change from 8 weeks of training to 4 weeks of detraining and change from 4 weeks of detraining to 8 weeks of detraining
  Rate of torque production during maximal isometric contractions
Strength of knee extensors and knee flexors | First evaluation, change from first evaluation to baseline, change from baseline to 8 weeks of training, change from 8 weeks of training to 4 weeks of detraining and change from 4 weeks of detraining to 8 weeks of detraining
  Maximal isometric strength
Strength of knee extensors and knee flexors | First evaluation, change from first evaluation to baseline, change from baseline to 8 weeks of training, change from 8 weeks of training to 4 weeks of detraining and change from 4 weeks of detraining to 8 weeks of detraining
  Maximal concentric strength
Strength of knee extensors and knee flexors | First evaluation, change from first evaluation to baseline, change from baseline to 8 weeks of training, change from 8 weeks of training to 4 weeks of detraining and change from 4 weeks of detraining to 8 weeks of detraining
  Maximal eccentric strength

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Research Laboratory, School of Physical Education, Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil